CLINICAL TRIAL: NCT00078494
Title: Phase I/II Trial of Latent Membrane Protein (LMP) - 2 Immunization for the Assessment of the Natural History and the Immunization-Induced Immunological Response in Patients at High Risk for Recurrence of Anaplastic Nasopharyngeal Cancer
Brief Title: Peptide Vaccine to Prevent Recurrence of Nasopharyngeal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040118; 04-CC-0118; NCT00112541 (obsolete NCT alias)
Record Dates: First submitted 2004-02-27; First posted 2004-03-01 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-05

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Immunization; Vaccine; Nasopharyngeal Cancer; Immunotherapy; Cancer; NPC
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Neoplasms | interventions — EBV-associated membrane antigen, Epstein-Barr virus

INTERVENTIONS:
Drug: EBV-LMP-2

SUMMARY:
This study will examine the effectiveness and side effects of an experimental vaccine to prevent recurrence of nasopharyngeal cancer. The likelihood of this cancer returning is higher in patients whose original lesion was large, whose cancer had spread to the adjacent lymph nodes, or who had surgery for metastatic disease (cancer that spread beyond the primary site). Nasopharyngeal tumors are caused by a common virus called Epstein-Barr virus, which produces a protein called LMP-2. Vaccination with specific pieces, or peptides, of the LMP-2 protein may boost the immune system's fight against the cancer. The vaccine injections are mixed with an oil-based substance called Montanide ISA-51, which is intended to increase the immune response to the peptide.

Patients 18 years of age and older whose nasopharyngeal cancer has been controlled by standard treatment with surgery, chemotherapy, or radiation therapy and who are currently free of disease may be eligible for this study. Candidates are screened with a physical examination and blood and urine tests. x-rays and other imaging studies are also done in patients who have not had these tests recently. All candidates are tested for HLA tissue type. Only patients with type HLA-A*1101 or HLA-A*2402 - the types on which the two vaccines in this study are based - receive vaccine therapy; others are offered standard medical treatment and observation.

Participants are randomly assigned to receive injections of one of two different vaccines (LMP-2:340-349 or LMP-2:419-427) to determine which peptide may offer the best immunity. Each treatment course consists of weekly immunizations for 8 consecutive weeks. The injections are given under the skin of the thigh. After every other treatment course (about every 3 months), patients undergo a series of x-rays and scans to look for tumor. The immunizations are given at the NIH Clinical Center. Patients are monitored for 1 hour after each injection and have blood tests and a physical examination to look for treatment side effects. Immunizations may continue for up to 12 months as long as the cancer does not return.

Patients are followed with blood tests every 12 weeks to monitor body functions. They also undergo leukapheresis-a procedure to collect white blood cells-before starting treatment and about 3 to 4 weeks after the fourth vaccine to evaluate how the vaccines affect the action of the immune system cells. For this procedure, blood is drawn through a needle in the arm, similar to donating blood. The blood is processed by a machine that separates and removes the lymphocytes (white blood cells), and the rest of the blood is returned through a needle in the other arm. Patients not receiving the vaccine also undergo leukapheresis to assess their natural response to LMP-2. Some patients may have a biopsy-surgical removal of a small piece of tissue under local anesthetic-of normal skin and tumor or lymph node tissue to examine the vaccine's effects on the tumor immune cells.

Patients who show no evidence of immunization against the LMP-2 protein after two courses of vaccine treatment are subsequently be followed with observation alone. Those who do respond to the vaccine are offered two additional courses of treatment to strengthen the response or to be followed by observation alone. Patients whose disease recurs after completing the first two treatment courses are taken off the study and referred back to their local physician or to another study, if an appropriate one is available.

DETAILED DESCRIPTION:
HLA-A*1101 and HLA-A*2402 positive patients with locally controlled anaplastic nasopharyngeal carcinoma at risk for loco-regional or distant recurrence will receive immunization with peptides representing HLA-restricted T cell epitopes of the Epstein-Barr virus encoded latent membrane protein-2 (LMP-2) emulsified in Montanide ISA-51. Patients will be allocated to treatment according to their HLA phenotype. The immunologic potential of the vaccine will be followed by enumerating the frequency of vaccines-specific CD8+ T cells in the peripheral blood using tetrameric HLA/peptide complexes. This study is designed to evaluate the immunologic effectiveness of peptide immunization in adjuvant settings in the context of anaplastic NPC.

ELIGIBILITY:
INCLUSION CRITERIA:

1. HLA-A*1101 and HLA-A*2402 patients, greater than 18 years of age, with advanced local disease (T3-T4N0-1M0), nodal disease (T1-T2N2-3M0) and loco-regional disease (T3-T4N2-3M0) at onset but presently controlled by standard therapy (combination of chemotherapy and radiotherapy) or with completely resected metastatic disease, 3 months after the completion of their primary treatment will be considered.

   All subjects will be judged disease free based on physical examination, ENT endoscopy, CT scan of abdomen, chest, neck and nasal sinuses and MRI of the head. All subjects must have received standard surgical, chemotherapy and radiation therapy appropriate for their stage of disease.

   Currently, standard treatment for locally advanced NPC in the U.S. consists of concomitant cisplatin with radiation followed by 3 courses of cisplatin and 5-fluorouracil. This, or comparable standard therapies will be considered part of standard therapy and patients will be considered for accrual three or more months after its completion. Patients must demonstrate evidence of local control with no histological or radiological evidence of recurrent disease three months after the end of standard therapy and be, otherwise, clinically disease free at the time of protocol entry as documented by radiological studies within 6 weeks of patient entry. Physical and histological evidence of disease recurrence at the time of patients' screening and during follow up will be performed under the supervision of Dr. Carter Van Waes during an out patient evaluation. Similar enrollment criteria will be used with patients who do not bear HLA-A*1101 or HLA-A*2402. However, these patients will be followed by observation only.
2. Pathologic confirmation of nasopharyngeal carcinoma by the NCI Laboratory of Pathology (NPC).
3. serum creatinine of 2.0 mg/dl or less,
4. Total bilirubin 1.6 mg/dl or less, except for patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
5. WBC 3000/mm(3) or greater,
6. platelet count 90,000 mm(3) or greater,
7. serum AST/ALT less than three times normal,
8. ECOG performance status of 0 or 1.
9. Patients of both genders must be willing to practice effective birth control during this trial because the potential for teratogenic effects are unknown.
10. Patients may have had prior adjuvant treatment or may have had treatment for metastatic disease and are now with no evidence of disease, including chemotherapy or biotherapy, as long as 1 month has elapsed since prior systemic therapy.

EXCLUSION CRITERIA:

Patients will be excluded:

1. Who are undergoing or have undergone in the past 3 weeks any systemic therapy except surgery for their cancer, and must have recovered from any adverse effects of treatment prior to entry, other than those that do not have clinical implications, e.g. alopecia. In the case a patient has received surgical intervention; at least one month should pass before enrollment in the study. All toxicity from previous therapy must have resolved to less than or equal to Grade 1 by NCI-CTC v 3.0 before enrollment.
2. Who have active systemic infections, autoimmune disease or any known immunodeficiency disease.

d. Who require systemic steroid therapy.

e. Who are pregnant (because of possible side effects on the fetus) or breastfeeding (because of unknown effects on the developing child).

f. Who are known to be positive for hepatitis BsAG or HIV antibody (because of possible immune effects of these conditions). Patients who may screen or have history positive for hepatitis C may be enrolled if their transaminases levels are within the limits specified in inclusion criteria.

g. Who have any form of active primary or secondary immunodeficiency or who have not recovered immune competence after chemotherapy or radiation therapy. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.) Active or secondary immunodeficiency will be judged based on the patient past medical history and normality of circulating T and B cell counts (Normal range 650-2, 108 and 49 to 424 respectively, Department of Laboratory Medicine, CC). In the similar fashion recovery from chemotherapy and radiation therapy will be evaluated. Previous experience in patients with melanoma or renal cell carcinoma who underwent chemotherapy of local radiation demonstrated that they immune response to common T cell epitopes such as Flu or Cytomegalovirus are rapidly restored within the first month from such treatment (unpublished observation).

h. Who have known hypersensitivity to any of the agents used in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99
Dates: Start 2004-02; Study Completion 2006-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenberg SA. Cancer vaccines based on the identification of genes encoding cancer regression antigens. Immunol Today. 1997 Apr;18(4):175-82. doi: 10.1016/s0167-5699(97)84664-6. No abstract available. PMID 9136454
- [Background] Boon T, Coulie PG, Van den Eynde B. Tumor antigens recognized by T cells. Immunol Today. 1997 Jun;18(6):267-8. doi: 10.1016/s0167-5699(97)80020-5. No abstract available. PMID 9190110
- [Background] Cormier JN, Salgaller ML, Prevette T, Barracchini KC, Rivoltini L, Restifo NP, Rosenberg SA, Marincola FM. Enhancement of cellular immunity in melanoma patients immunized with a peptide from MART-1/Melan A. Cancer J Sci Am. 1997 Jan-Feb;3(1):37-44. PMID 9072306